CLINICAL TRIAL: NCT02660450
Title: Relationship Between Methods of Aerobic Prescription: Heart Rate vs. VO2 Load vs. Self Selected
Brief Title: Relationship Between Aerobic Prescription Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Alberto Souza de Sá Filho, Doctorade in Mental Health, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: UNIG 02
Record Dates: First submitted 2016-01-04; First posted 2016-01-21 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
MeSH Terms: interventions — Prescriptions; Workload; Heart Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Prescription for Workload (Experimental): Prescription from 65% VO2max for 5 min of exercise
  Interventions: Other: Prescription for Heart Rate; Other: Prescription Self Selected
- Prescription for Heart Rate (Experimental): Prescription from 60 - 65% Maximum Heart Rate for 5 min of exercise
  Interventions: Other: Prescription for Workload; Other: Prescription Self Selected
- Prescription Self Selected (Experimental): Prescription Self Selected from Perceived exertion at 3 - 4 (moderate) for 5 min of exercise
  Interventions: Other: Prescription for Workload; Other: Prescription for Heart Rate

INTERVENTIONS:
Other: Prescription for Workload — Prescription from 65% VO2max for 5 min of exercise
  Other Names: VO2Max
  Arms: Prescription Self Selected; Prescription for Heart Rate
Other: Prescription for Heart Rate — Prescription from 60 - 65% Maximum Heart Rate for 5 min of exercise
  Other Names: Heart Rate
  Arms: Prescription Self Selected; Prescription for Workload
Other: Prescription Self Selected — Prescription Self Selected from Perceived exertion at 3 - 4 (moderate) for 5 min of exercise
  Other Names: Self Selected
  Arms: Prescription for Heart Rate; Prescription for Workload

SUMMARY:
Current literature report 3 ways to prescribe and control aerobic training. Such models require comparison to determine if they really provide the same impact training in a prescription. The aim of this study is to compare the results of different methods of prescription of aerobic training, ie VO2 workload, heart rate (HR), and load self adjusted by perceived effort (PSE) as well as psychological responses activation, and feel depending on the stimuli offered.

DETAILED DESCRIPTION:
36 subjects will undergo two sessions. On the first visit, a maximum aerobic exercise test will be carried on treadmill to determine the maximum oxygen intake and maximum heart rate. Second, the subjects are placed (in a blinded fashion) in 3 situations of moderate effort (60 to 65%) for a total of 5 min and 3 min interval between conditions. In situation 1) will be used to speed regarding the particular metabolic demand from the maximum oxygen intake; In the second situation the reserve of heart rate will be used as reference for prescription aiming to achieve 60-65%; On the last visit will be shown to subjects a perceived effort characterized as moderate and asked to adjust their speed according to the application effort. The final will be recorded each time the FC and the speed and perception of effort that the subject was.

ELIGIBILITY:
Inclusion Criteria:

* 18 at 45 years
* Risk stratification low
* Physically active by American College of Sports Medicine criteria

Exclusion Criteria:

* Use of ergogenic resources
* Use of sympatholytic drugs
* Use of stimulants

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-04 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Response of Heart Rate and perceived Effort through prescriptions for oxygen uptake | Acute Change in 5 minutes of moderate aerobic exercise
Response of Heart Rate through prescriptions for self selected workload based in perceived effort | Acute Change in 5 minutes of moderate aerobic exercise
Response of velocity and Perceived Effort through Prescription of Heart Rate | Acute Change in 5 minutes of moderate aerobic exercise

IPD SHARING:
Plan to Share IPD: Undecided